CLINICAL TRIAL: NCT02890992
Title: An 8-Week Open-Label, Sequential, Repeated Dose-Finding Study to Evaluate the Efficacy and Safety of Alirocumab in Children and Adolescents With Heterozygous Familial Hypercholesterolemia Followed by an Extension Phase
Brief Title: An 8-Week Dose-Finding Study to Evaluate the Efficacy and Safety of Alirocumab in Children and Adolescents With Heterozygous Familial Hypercholesterolemia
Acronym: ODYSSEY KIDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DFI14223; 2015-003766-85 (EudraCT Number); U1111-1178-4764 (Other: UTN)
Record Dates: First submitted 2016-08-31; First posted 2016-09-07 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-08

CONDITIONS: Hypercholesterolaemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Ezetimibe; Cholestyramine Resin; Fenofibrate; Fatty Acids, Omega-3; Niacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Cohort 1 - Alirocumab 30 mg Q2W: <50 kg (Experimental): Period 1: Participants with body weight less than (<) 50 kilograms (kg) received subcutaneous (SC) injection of alirocumab 30 milligram(mg) administered every 2 weeks (Q2W) up to 8 weeks added to lipid modifying therapy (LMT).
  Period 2: Participants with body weight < 50 kg received SC injection of alirocumab 30 mg administered Q2W from Week 16 until they started receiving dose matching to Cohort 2 dosage including dose adjustment to body weight as required. Cohort 2 dosage was: if body weight was still < 50 kg, participants received SC injection of alirocumab 40 mg administered Q2W until Week 130; if body weight was > = 50 kg participants received SC injection of alirocumab 75 mg administered Q2W until Week 130.
  Interventions: Drug: alirocumab SAR236553 (REGN727); Drug: statins; Drug: ezetimibe; Drug: cholestyramine; Drug: fenofibrate; Drug: omega-3 fatty acids; Drug: nicotinic acid
- Cohort 1 - Alirocumab 50 mg Q2W: >=50 kg (Experimental): Period 1: Participants with body weight greater than or equal to (>=) 50 kg received SC injection of alirocumab 50 mg administered Q2W up to 8 weeks added to LMT.
  Period 2: Participants with body weight >= 50 kg received SC injection of alirocumab 50 mg administered Q2W from Week 16 until switch to Cohort 2 dosage then SC injection of alirocumab 75 mg administered Q2W until Week 130.
  Interventions: Drug: alirocumab SAR236553 (REGN727); Drug: statins; Drug: ezetimibe; Drug: cholestyramine; Drug: fenofibrate; Drug: omega-3 fatty acids; Drug: nicotinic acid
- Cohort 2 - Alirocumab 40 mg Q2W: <50 kg (Experimental): Period 1: Participants with body weight < 50 kg received SC injection of alirocumab 40 mg administered Q2W up to 8 weeks added to LMT.
  Period 2: Participants with body weight < 50 kg received SC injection of alirocumab 40 mg administered Q2W from Week 16 until switch of dosage in Cohorts 1 and 3. If body weight was still < 50 kg, participants continued to receive SC injection of alirocumab 40 mg administered Q2W until Week 130; if body weight was > = 50 kg participants received SC injection of alirocumab 75 mg administered Q2W until Week 130.
  Interventions: Drug: alirocumab SAR236553 (REGN727); Drug: statins; Drug: ezetimibe; Drug: cholestyramine; Drug: fenofibrate; Drug: omega-3 fatty acids; Drug: nicotinic acid
- Cohort 2 - Alirocumab 75 mg Q2W: >=50 kg (Experimental): Period 1: Participants with body weight >= 50 kg received SC injection of alirocumab 75 mg administered Q2W up to 8 weeks added to LMT.
  Period 2: Participants with body weight >= 50 kg received SC injection of alirocumab 75 mg administered Q2W from Week 16 until Week 130.
  Interventions: Drug: alirocumab SAR236553 (REGN727); Drug: statins; Drug: ezetimibe; Drug: cholestyramine; Drug: fenofibrate; Drug: omega-3 fatty acids; Drug: nicotinic acid
- Cohort 3 - Alirocumab 75 mg Q4W: <50 kg (Experimental): Period 1: Participants with body weight < 50 kg received SC injection of alirocumab 75 mg administered every 4 weeks (Q4W) up to 8 weeks added to LMT.
  Period 2: Participants with body weight < 50 kg received SC injection of alirocumab 75 mg administered Q4W from Week 14 until switch to Cohort 2 dosage including dose adjustment to body weight as required, then Cohort 2 dosage: if body weight was still < 50 kg, participants received SC injection of alirocumab 40 mg administered Q2W until Week 130; if body weight was > = 50 kg participants received SC injection of alirocumab 75 mg administered Q2W until Week 130.
  Interventions: Drug: alirocumab SAR236553 (REGN727); Drug: statins; Drug: ezetimibe; Drug: cholestyramine; Drug: fenofibrate; Drug: omega-3 fatty acids; Drug: nicotinic acid
- Cohort 3 - Alirocumab 150 mg Q4W: >=50 kg (Experimental): Period 1: Participants with body weight >= 50 kg received SC injection of alirocumab 150 mg administered Q4W up to Week 8 added to LMT.
  Period 2: Participants with body weight >= 50 kg received SC injection of alirocumab 150 mg administered Q4W from Week 14 until switch to Cohort 2 dosage then SC injection of alirocumab 75 mg administered Q2W until Week 130.
  Interventions: Drug: alirocumab SAR236553 (REGN727); Drug: statins; Drug: ezetimibe; Drug: cholestyramine; Drug: fenofibrate; Drug: omega-3 fatty acids; Drug: nicotinic acid
- Cohort 4 - Alirocumab 150 mg Q4W: <50 kg (Experimental): Period 1: Participants with body weight < 50 kg received SC injection of alirocumab 150 mg administered Q4W up to 12 weeks added to LMT.
  Period 2: Participants with body weight < 50 kg received SC injection of Alirocumab 150 mg administered Q4W from Week 12 until Week 48.
  Interventions: Drug: alirocumab SAR236553 (REGN727); Drug: statins; Drug: ezetimibe; Drug: cholestyramine; Drug: fenofibrate; Drug: omega-3 fatty acids; Drug: nicotinic acid
- Cohort 4 - Alirocumab 300 mg Q4W: >=50 kg (Experimental): Period 1: Participants with body weight >= 50 kg received SC injection of alirocumab 300 mg administered Q4W up to 12 weeks added to LMT.
  Period 2: Participants with body weight >= 50 kg received SC injection of alirocumab 300 mg administered Q4W from Week 12 until Week 48.
  Interventions: Drug: alirocumab SAR236553 (REGN727); Drug: statins; Drug: ezetimibe; Drug: cholestyramine; Drug: fenofibrate; Drug: omega-3 fatty acids; Drug: nicotinic acid

INTERVENTIONS:
Drug: alirocumab SAR236553 (REGN727) — Pharmaceutical form: solution Route of administration: subcutaneous injection
  Other Names: Praluent
Drug: statins — Pharmaceutical form: tablet Route of administration: oral
Drug: ezetimibe — Pharmaceutical form:tablet Route of administration: oral
Drug: cholestyramine — Pharmaceutical form:tablet Route of administration: oral
Drug: fenofibrate — Pharmaceutical form: tablet Route of administration: oral
Drug: omega-3 fatty acids — Pharmaceutical form: tablet Route of administration: oral
Drug: nicotinic acid — Pharmaceutical form: tablet Route of administration: oral

SUMMARY:
Primary Objective:

To evaluate the effect of alirocumab on low-density lipoprotein cholesterol (LDL-C) levels after 8 weeks of treatment in heterozygous familial hypercholesterolemia (heFH) participants aged of 8 to 17 years, with LDL-C >=130 milligrams per deciliter (mg/dL) (3.37 millimoles per litre [mmol/L]) on optimal stable daily dose of statin therapy +/- other lipid modifying therapies (LMTs) or a stable dose of non-statin LMTs in case of intolerance to statins for at least 4 weeks prior to the screening period.

Secondary Objective:

* To evaluate the safety and tolerability of alirocumab.
* To evaluate the pharmacokinetics profile of alirocumab.
* To evaluate the effects of alirocumab on other lipid parameters.

DETAILED DESCRIPTION:
For Cohorts 1 to 3, a study duration of approximately 16-23 weeks (screening period: up to 6 (+1) weeks, open-label dose finding treatment period: 8 weeks, follow up period: 6-8 weeks).

For Cohort 4, a study duration of approximately 14-19 weeks (screening period up to 6 [+1] weeks, open-label dose finding treatment period: 12 weeks).

Optional extension period: up to a maximum of 2 years for the first participants enrolled in Cohorts 1 to 3, but a maximum of approximately 5 months for the first participants enrolled in Cohort 4.

For all participants who declined participation in the phase 3 study, their last alirocumab injection was on December 2018.

ELIGIBILITY:
Inclusion criteria :

* Children and adolescent male and female participants aged of 8 to 17 years at the time of signed informed consent. For Russia only: Male and female participants aged >=12 and <=17 years at the time of signed informed consent.
* Participants with diagnosis of heterozygous familial hypercholesterolemia (heFH) through genotyping or clinical criteria.
* Participants treated with optimal dose of statin +/- other LMT(s) or non-statin LMT(s) if statin intolerant at stable dose for at least 4 weeks prior to screening lipid sampling.
* Participants with calculated LDL-C greater than or equal to 130 mg/dL (>=3.37 mmol/L) at the screening visit.
* Participants with body weight greater than or equal to 25 kg.
* Participants aged of 8 to 9 years to be at Tanner stage 1 and participants aged of 10 to 17 years to be at least at Tanner stage 2 in their development.
* A signed informed consent indicating parental permission with or without participant assent.

Exclusion criteria:

* Participant with secondary hyperlipidemia.
* Diagnosis of homozygous familial hypercholesterolemia.
* Participant who had received lipid apheresis treatment within 2 months prior to the screening period, or has plans to receive it during the study.
* Known history of type 1 or type 2 diabetes mellitus.
* Known history of thyroid disease.
* Known history of hypertension.
* Fasting triglycerides >350 mg/dL (3.95 mmol/L).
* Severe renal impairment (i.e., estimated glomerular filtration rate [eGFR] <30 mL/min/1.73 m^2).
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2 x upper limit of normal (ULN).
* Creatinine phosphokinase (CPK) >3 x ULN.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2018-09-13 (Actual); Study Completion 2019-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (16):
- United States (3):
  - Investigational Site Number 8400002, St Louis, Missouri
  - Investigational Site Number 8400005, Charlotte, North Carolina
  - Investigational Site Number 8400001, Cincinnati, Ohio
- Investigational Site Number 1240001, Québec, Canada
- Czechia (3):
  - Investigational Site Number 2030001, Brno
  - Investigational Site Number 2030003, Praha 5 - Motol
  - Investigational Site Number 2030002, Zlín
- Investigational Site Number 2500001, Bron, France
- Investigational Site Number 5280001, Amsterdam, Netherlands
- Investigational Site Number 5780001, Oslo, Norway
- Russia (2):
  - Investigational Site Number 6430001, Kemerovo
  - Investigational Site Number 6430004, Saint Petersburg
- Investigational Site Number 7100001, Parow, South Africa
- Spain (2):
  - Investigational Site Number 7240004, A Coruña
  - Investigational Site Number 7240001, Madrid
- Investigational Site Number 7520001, Stockholm, Sweden

REFERENCES:
- [Derived] Daniels S, Caprio S, Chaudhari U, Manvelian G, Baccara-Dinet MT, Brunet A, Scemama M, Loizeau V, Bruckert E. PCSK9 inhibition with alirocumab in pediatric patients with heterozygous familial hypercholesterolemia: The ODYSSEY KIDS study. J Clin Lipidol. 2020 May-Jun;14(3):322-330.e5. doi: 10.1016/j.jacl.2020.03.001. Epub 2020 Mar 28. PMID 32331936

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 16 sites in 10 countries. Overall 63 participants were screened between 15 September 2016 and 13 June 2018, of whom 21 participants were screen failures. Screen failures were mainly due to exclusion criteria met.
Pre-assignment Details: A total of 42 participants were included in this study.
Groups:
- Cohort 1 - Alirocumab 30 mg Q2W: <50 kg: Period 1: Participants with body weight less than (<) 50 kilograms (kg) received subcutaneous (SC) injection of alirocumab 30 milligram (mg) administered every 2 weeks (Q2W) up to 8 weeks added to lipid modifying therapy (LMT).
  Period 2: Participants with body weight < 50 kg received SC injection of alirocumab 30 mg administered Q2W from Week 16 until switch to Cohort 2 dosage including dose adjustment to body weight as required, then Cohort 2 dosage: if body weight was still < 50 kg, participants received SC injection of alirocumab 40 mg administered Q2W until Week 130; if body weight was > = 50 kg participants received SC injection of alirocumab 75 mg administered Q2W until Week 130.
- Cohort 3 - Alirocumab 75 mg Q4W: <50 kg: Period 1: Participants with body weight < 50 kg received SC injection of alirocumab 75 mg administered Q4W up to 8 weeks added to LMT.
  Period 2: Participants with body weight < 50 kg received SC injection of alirocumab 75 mg administered Q4W from Week 14 until switch to Cohort 2 dosage including dose adjustment to body weight as required, then Cohort 2 dosage: if body weight was still < 50 kg, participants received SC injection of alirocumab 40 mg administered Q2W until Week 130; if body weight was > = 50 kg participants received SC injection of alirocumab 75 mg administered Q2W until Week 130.
Period: 12 Weeks Open-Label Dose Finding Period
Arm/Group | Cohort 1 - Alirocumab 30 mg Q2W: <50 kg | Cohort 1 - Alirocumab 50 mg Q2W: >=50 kg | Cohort 2 - Alirocumab 40 mg Q2W: <50 kg | Cohort 2 - Alirocumab 75 mg Q2W: >=50 kg | Cohort 3 - Alirocumab 75 mg Q4W: <50 kg | Cohort 3 - Alirocumab 150 mg Q4W: >=50 kg | Cohort 4 - Alirocumab 150 mg Q4W: <50 kg | Cohort 4 - Alirocumab 300 mg Q4W: >=50 kg
Started | 4 | 6 | 4 | 6 | 6 | 5 | 6 | 5
Treated | 4 | 6 | 4 | 6 | 6 | 5 | 6 | 5
Completed | 4 (Out of 4 participants, 3 participants entered into the open-label extension (OLE) period.) | 6 | 4 | 6 | 6 | 5 | 6 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: 130 Weeks Open-Label Extension Period
Arm/Group | Cohort 1 - Alirocumab 30 mg Q2W: <50 kg | Cohort 1 - Alirocumab 50 mg Q2W: >=50 kg | Cohort 2 - Alirocumab 40 mg Q2W: <50 kg | Cohort 2 - Alirocumab 75 mg Q2W: >=50 kg | Cohort 3 - Alirocumab 75 mg Q4W: <50 kg | Cohort 3 - Alirocumab 150 mg Q4W: >=50 kg | Cohort 4 - Alirocumab 150 mg Q4W: <50 kg | Cohort 4 - Alirocumab 300 mg Q4W: >=50 kg
Started | 3 (3 participants from Open-Label Dose Finding Period (OLDFI) entered in OLE period.) | 6 | 4 | 6 | 6 | 5 | 6 | 5
Treated | 3 | 6 | 4 | 6 | 6 | 5 | 5 | 4
Completed | 3 | 3 | 4 | 6 | 6 | 5 | 5 | 4
Not Completed | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Included but not treated | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Other than specified | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on safety population that included population who did actually received at least one dose or part of a dose of the open-label investigational medicinal product (IMP). Participants were analyzed according to the dose of alirocumab actually received.
Groups:
- Cohort 1 - Alirocumab 30 mg Q2W: <50 kg: Period 1: Participants with body weight < 50 kg received SC injection of alirocumab 30 mg administered Q2W up to 8 weeks added to LMT.
  Period 2: Participants with body weight < 50 kg received SC injection of alirocumab 30 mg administered Q2W from Week 16 until switch to Cohort 2 dosage including dose adjustment to body weight as required, then Cohort 2 dosage: if body weight was still < 50 kg, participants received SC injection of alirocumab 40 mg administered Q2W until Week 130; if body weight was > = 50 kg participants received SC injection of alirocumab 75 mg administered Q2W until Week 130.
- Cohort 1 - Alirocumab 50 mg Q2W: >=50 kg: Period 1: Participants with body weight >= 50 kg received SC injection of alirocumab 50 mg administered Q2W up to 8 weeks added to LMT.
  Period 2: Participants with body weight >= 50 kg received SC injection of alirocumab 50 mg administered Q2W from Week 16 until switch to Cohort 2 dosage then SC injection of alirocumab 75 mg administered Q2W until Week 130.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - Alirocumab 30 mg Q2W: <50 kg | Cohort 1 - Alirocumab 50 mg Q2W: >=50 kg | Cohort 2 - Alirocumab 40 mg Q2W: <50 kg | Cohort 2 - Alirocumab 75 mg Q2W: >=50 kg | Cohort 3 - Alirocumab 75 mg Q4W: <50 kg | Cohort 3 - Alirocumab 150 mg Q4W: >=50 kg | Cohort 4 - Alirocumab 150 mg Q4W: <50 kg | Cohort 4 - Alirocumab 300 mg Q4W: >=50 kg | Total
Number analyzed (Participants) | 4 | 6 | 4 | 6 | 6 | 5 | 6 | 5 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.0 (2.0) | 13.8 (2.7) | 11.3 (2.2) | 14.3 (2.3) | 9.8 (1.9) | 13.8 (1.6) | 11.3 (2.2) | 13.6 (2.1) | 12.4 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 2 | 2 | 3 | 3 | 1 | 2 | 19
  Male | 2 | 2 | 2 | 4 | 3 | 2 | 5 | 3 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Black or African American/White | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  White | 4 | 6 | 4 | 6 | 5 | 5 | 6 | 3 | 39
Low Density Lipoprotein Cholesterol (LDL-C) [Mean (Standard Deviation); unit: millimoles per litre (mmol/L)] | 5.169 (0.736) | 4.339 (1.200) | 3.596 (0.630) | 4.510 (1.052) | 4.337 (1.147) | 4.642 (1.272) | 5.100 (1.136) | 4.641 (0.926) | 4.6 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Calculated Low Density Lipoprotein Cholesterol (LDL-C) at Week 8
Description: Percent change in calculated LDL-C was defined as 100*(calculated LDL-C value at Week 8 - calculated LDL-C value at baseline)/calculated LDL-C value at baseline. All available baseline and post-baseline calculated LDL-C value during the OLDFI efficacy treatment period & within one of the analysis windows up to Week 8 were used in the model. OLDFI efficacy treatment period was defined as the period from first investigational medicinal product (IMP) injection to last OLDFI IMP injection + 21 days(for Cohorts 1 & 2) or +35 days (for Cohorts 3 & 4). Adjusted Least-squares (LS) mean & standard error (SE) at Week 8 were obtained from mixed-effect model with repeated measures (MMRM) analysis, with fixed categorical effects of alirocumab dose/dose regimen (30 mg Q2W [<50 kg], 40 mg Q2W [<50 kg], 50 mg Q2W [>=50 kg], 75 mg Q2W [>=50 kg], 75 mg Q4W [<50 kg],150 mg Q4W [>=50 kg], 150 mg Q4W [<50 kg] and 300 mg Q4W ([>=50 kg] dose), time point & dose/dose regimen-by-time point interaction.
Time Frame: Baseline, Week 8
Population: Analysis was performed on modified intent-to-treat (mITT) population which included all participants who received at least one dose or partial dose of IMP injection and had an evaluable outcome measure during the open-label dose finding efficacy treatment period.
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- Cohort 1 - Alirocumab 30 mg Q2W: <50 kg: Participants with body weight < 50 kg received SC injection of alirocumab 30 mg administered Q2W up to 8 weeks added to LMT.
- Cohort 1 - Alirocumab 50 mg Q2W: >=50 kg: Participants with body weight >= 50 kg received SC injection of alirocumab 50 mg administered Q2W up to 8 weeks added to LMT.
- Cohort 2 - Alirocumab 40 mg Q2W: <50 kg: Participants with body weight < 50 kg received SC injection of alirocumab 40 mg administered Q2W up to 8 weeks added to LMT.
- Cohort 2 - Alirocumab 75 mg Q2W: >=50 kg: Participants with body weight >= 50 kg received SC injection of alirocumab 75 mg administered Q2W up to 8 weeks added to LMT.
- Cohort 3 - Alirocumab 75 mg Q4W: <50 kg: Participants with body weight < 50 kg received SC injection of alirocumab 75 mg administered Q4W up to 8 weeks added to LMT.
- Cohort 3 - Alirocumab 150 mg Q4W: >=50 kg: Participants with body weight >= 50 kg received SC injection of alirocumab 150 mg administered Q4W up to Week 8 added to LMT.
- Cohort 4 - Alirocumab 150 mg Q4W: <50 kg: Participants with body weight < 50 kg received SC injection of alirocumab 150 mg administered Q4W up to 12 weeks added to LMT.
- Cohort 4 - Alirocumab 300 mg Q4W: >=50 kg: Participants with body weight >= 50 kg received SC injection of alirocumab 300 mg administered Q4W up to 12 weeks added to LMT.
Arm/Group | Cohort 1 - Alirocumab 30 mg Q2W: <50 kg | Cohort 1 - Alirocumab 50 mg Q2W: >=50 kg | Cohort 2 - Alirocumab 40 mg Q2W: <50 kg | Cohort 2 - Alirocumab 75 mg Q2W: >=50 kg | Cohort 3 - Alirocumab 75 mg Q4W: <50 kg | Cohort 3 - Alirocumab 150 mg Q4W: >=50 kg | Cohort 4 - Alirocumab 150 mg Q4W: <50 kg | Cohort 4 - Alirocumab 300 mg Q4W: >=50 kg
Number analyzed (Participants) | 4 | 6 | 4 | 6 | 6 | 5 | 6 | 5
percent change | -41.1 (12.6) | -7.9 (10.3) | -40.6 (13.2) | -49.8 (10.6) | -17.5 (10.3) | 4.0 (11.2) | -31.9 (10.3) | -59.8 (11.2)

2. Secondary Outcome: Absolute Change From Baseline in Calculated Low Density Lipoprotein Cholesterol (LDL-C) at Week 8
Description: Absolute change in LDL-C was calculated by subtracting baseline value from Week 8 value. Adjusted LS means and SE were obtained using MMRM analysis, with fixed categorical effects of alirocumab dose/dose regimen, time point and dose/dose regimen-by-time point interaction.
Time Frame: Baseline, Week 8
Population: Analysis was performed on mITT population.
Measure: Least Squares Mean (Standard Error); unit: milligram per deciliter (mg/dL)
Groups:
- Cohort 1 - Alirocumab 30 mg Q2W: <50 kg: Participants with body weight < 50 kg received SC injection of alirocumab 30 milligram(mg) administered Q2W up to 8 weeks added to LMT.
Arm/Group | Cohort 1 - Alirocumab 30 mg Q2W: <50 kg | Cohort 1 - Alirocumab 50 mg Q2W: >=50 kg | Cohort 2 - Alirocumab 40 mg Q2W: <50 kg | Cohort 2 - Alirocumab 75 mg Q2W: >=50 kg | Cohort 3 - Alirocumab 75 mg Q4W: <50 kg | Cohort 3 - Alirocumab 150 mg Q4W: >=50 kg | Cohort 4 - Alirocumab 150 mg Q4W: <50 kg | Cohort 4 - Alirocumab 300 mg Q4W: >=50 kg
Number analyzed (Participants) | 4 | 6 | 4 | 6 | 6 | 5 | 6 | 5
milligram per deciliter (mg/dL) | -83.7 (19.5) | -27.6 (15.9) | -55.5 (20.8) | -88.3 (16.5) | -32.4 (15.9) | 0.1 (17.4) | -55.9 (15.9) | -104.3 (17.4)

3. Secondary Outcome: Percentage of Participants Achieving Calculated Low Density Lipoprotein Cholesterol (LDL-C) <130 mg/dL (3.37 mmol/L) at Week 8
Description: Combined estimate for percentage of participants was obtained by averaging out all the imputed percentage of participants reaching the level of interest. A two-step multiple imputation procedure was used to address missing values in the mITT population in the two steps respectively; with number of imputations = 1000. In the first step, the monotone missing pattern was induced in the multiply-imputed data. In the second step, the missing data at subsequent visits were imputed using the regression method for continuous variables.
Time Frame: At Week 8
Population: Analysis was performed on mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 - Alirocumab 30 mg Q2W: <50 kg | Cohort 1 - Alirocumab 50 mg Q2W: >=50 kg | Cohort 2 - Alirocumab 40 mg Q2W: <50 kg | Cohort 2 - Alirocumab 75 mg Q2W: >=50 kg | Cohort 3 - Alirocumab 75 mg Q4W: <50 kg | Cohort 3 - Alirocumab 150 mg Q4W: >=50 kg | Cohort 4 - Alirocumab 150 mg Q4W: <50 kg | Cohort 4 - Alirocumab 300 mg Q4W: >=50 kg
Number analyzed (Participants) | 4 | 6 | 4 | 6 | 6 | 5 | 6 | 5
percentage of participants | 100.0 | 33.3 | 97.6 | 83.0 | 33.3 | 20.0 | 66.7 | 80.0

4. Secondary Outcome: Percentage of Participants Achieving Calculated LDL-C <110 mg/dL (2.84 mmol/L) at Week 8
Description: as for outcome 3
Time Frame: At Week 8
Population: Analysis was performed on mITT population.
Measure: Number; unit: percentage of participants
Groups:
- Cohort 1 - Alirocumab 30 mg Q2W: <50 kg: Participants with body weight < 50 kg received SC injection of alirocumab 30 milligram (mg) administered Q2W up to 8 weeks added to LMT.
Arm/Group | Cohort 1 - Alirocumab 30 mg Q2W: <50 kg | Cohort 1 - Alirocumab 50 mg Q2W: >=50 kg | Cohort 2 - Alirocumab 40 mg Q2W: <50 kg | Cohort 2 - Alirocumab 75 mg Q2W: >=50 kg | Cohort 3 - Alirocumab 75 mg Q4W: <50 kg | Cohort 3 - Alirocumab 150 mg Q4W: >=50 kg | Cohort 4 - Alirocumab 150 mg Q4W: <50 kg | Cohort 4 - Alirocumab 300 mg Q4W: >=50 kg
Number analyzed (Participants) | 4 | 6 | 4 | 6 | 6 | 5 | 6 | 5
percentage of participants | 0.0 | 0.0 | 93.4 | 65.7 | 16.7 | 20.0 | 66.7 | 80.0

5. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 12: Cohort 4
Description: Adjusted LS means and standard error at Week 12 were obtained from MMRM analysis, with fixed categorical effects of alirocumab dose/dose regimen, time point and dose/dose regimen-by-time point interaction.
Time Frame: Baseline, Week 12
Population: Analysis was performed on mITT population. Data for this outcome measure was planned to be collected for Cohort 4 only.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Cohort 4 - Alirocumab 150 mg Q4W: <50 kg | Cohort 4 - Alirocumab 300 mg Q4W: >=50 kg
Number analyzed (Participants) | 6 | 5
percent change | -29.7 (6.9) | -49.2 (7.5)

6. Secondary Outcome: Percent Change From Baseline in Apolipoprotein (Apo) B at Week 8
Description: Adjusted LS means and SE at Week 8 were obtained from MMRM analysis, with fixed categorical effects of alirocumab dose/dose regimen, time point and dose/dose regimen-by-time point interaction. All available baseline value and post-baseline values in at least one of the analysis windows used in the model.
Time Frame: Baseline, Week 8
Population: Analysis was performed on mITT population. Here, overall number of participants analyzed=participants with available data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Cohort 1 - Alirocumab 30 mg Q2W: <50 kg | Cohort 1 - Alirocumab 50 mg Q2W: >=50 kg | Cohort 2 - Alirocumab 40 mg Q2W: <50 kg | Cohort 2 - Alirocumab 75 mg Q2W: >=50 kg | Cohort 3 - Alirocumab 75 mg Q4W: <50 kg | Cohort 3 - Alirocumab 150 mg Q4W: >=50 kg | Cohort 4 - Alirocumab 150 mg Q4W: <50 kg | Cohort 4 - Alirocumab 300 mg Q4W: >=50 kg
Number analyzed (Participants) | 3 | 6 | 3 | 6 | 6 | 5 | 6 | 5
percent change | -38.4 (12.8) | -9.7 (9.1) | -36.4 (12.8) | -40.1 (9.9) | -12.6 (9.1) | -0.9 (9.9) | -27.2 (9.1) | -51.4 (9.9)

7. Secondary Outcome: Percent Change From Baseline in Non-High Density Lipoprotein (HDL-C) at Week 8
Description: Adjusted LS means and SE at Week 8 were obtained from MMRM analysis, with fixed categorical effects of alirocumab dose/dose regimen, time point and dose/dose regimen-by-time point interaction. All available baselines value and post-baseline values in at least one of the analysis windows up to Week 8 were used in the model.
Time Frame: Baseline, Week 8
Population: Analysis was performed on mITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Cohort 1 - Alirocumab 30 mg Q2W: <50 kg | Cohort 1 - Alirocumab 50 mg Q2W: >=50 kg | Cohort 2 - Alirocumab 40 mg Q2W: <50 kg | Cohort 2 - Alirocumab 75 mg Q2W: >=50 kg | Cohort 3 - Alirocumab 75 mg Q4W: <50 kg | Cohort 3 - Alirocumab 150 mg Q4W: >=50 kg | Cohort 4 - Alirocumab 150 mg Q4W: <50 kg | Cohort 4 - Alirocumab 300 mg Q4W: >=50 kg
Number analyzed (Participants) | 4 | 6 | 4 | 6 | 6 | 5 | 6 | 5
percent change | -39.6 (11.9) | -7.1 (9.7) | -39.7 (12.5) | -43.9 (10.0) | -14.4 (9.7) | 3.2 (10.7) | -31.5 (9.7) | -54.6 (10.7)

8. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (Total-C) at Week 8
Description: Adjusted LS means and SE at Week 8 were obtained from MMRM analysis, with fixed categorical effects of alirocumab dose/dose regimen, time point and dose/dose regimen-by-time point interaction. All available baseline values and post-baseline values in at least one of the analysis windows up to Week 8 were used in the model.
Time Frame: Baseline, Week 8
Population: Analysis was performed on mITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Cohort 1 - Alirocumab 30 mg Q2W: <50 kg | Cohort 1 - Alirocumab 50 mg Q2W: >=50 kg | Cohort 2 - Alirocumab 40 mg Q2W: <50 kg | Cohort 2 - Alirocumab 75 mg Q2W: >=50 kg | Cohort 3 - Alirocumab 75 mg Q4W: <50 kg | Cohort 3 - Alirocumab 150 mg Q4W: >=50 kg | Cohort 4 - Alirocumab 150 mg Q4W: <50 kg | Cohort 4 - Alirocumab 300 mg Q4W: >=50 kg
Number analyzed (Participants) | 4 | 6 | 4 | 6 | 6 | 5 | 6 | 5
percent change | -29.0 (9.7) | -4.1 (7.9) | -28.6 (10.1) | -34.2 (8.1) | -10.7 (7.9) | 5.2 (8.6) | -24.0 (7.9) | -41.8 (8.6)

9. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a) at Week 8
Description: Combined estimates and SE were obtained by combining adjusted means and SE from robust regression model analyses of the different imputed data sets. The robust regression models included the fixed categorical effect of alirocumab dose/dose regimen. A two-step multiple imputation procedure was used to address missing values in the mITT population in the two steps respectively (with number of imputations = 1000). In the first step, the monotone missing pattern was induced in the multiply-imputed data. In the second step, the missing data at subsequent visits were imputed using the regression method for continuous variables.
Time Frame: Baseline, Week 8
Population: Analysis was performed on mITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Cohort 1 - Alirocumab 30 mg Q2W: <50 kg | Cohort 1 - Alirocumab 50 mg Q2W: >=50 kg | Cohort 2 - Alirocumab 40 mg Q2W: <50 kg | Cohort 2 - Alirocumab 75 mg Q2W: >=50 kg | Cohort 3 - Alirocumab 75 mg Q4W: <50 kg | Cohort 3 - Alirocumab 150 mg Q4W: >=50 kg | Cohort 4 - Alirocumab 150 mg Q4W: <50 kg | Cohort 4 - Alirocumab 300 mg Q4W: >=50 kg
Number analyzed (Participants) | 4 | 6 | 4 | 6 | 6 | 5 | 6 | 5
percent change | 4.5 (21.1) | -26.9 (11.6) | 1.5 (15.1) | -25.2 (14.4) | 2.2 (10.5) | -7.7 (11.4) | 0.1 (10.2) | -7.7 (11.1)

10. Secondary Outcome: Percent Change From Baseline in Fasting Triglyceride at Week 8
Description: Combined estimates and SE were obtained by combining adjusted means and SE from robust regression model analyses of the different imputed data sets. The robust regression models included the fixed categorical effect of alirocumab dose/dose regimen. A two-step multiple imputation procedure was used to address missing values in the mITT population (in the two steps respectively; with number of imputations = 1000). In the first step, the monotone missing pattern was induced in the multiply-imputed data. In the second step, the missing data at subsequent visits were imputed using the regression method for continuous variables.
Time Frame: Baseline, Week 8
Population: Analysis was performed on mITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Cohort 1 - Alirocumab 30 mg Q2W: <50 kg | Cohort 1 - Alirocumab 50 mg Q2W: >=50 kg | Cohort 2 - Alirocumab 40 mg Q2W: <50 kg | Cohort 2 - Alirocumab 75 mg Q2W: >=50 kg | Cohort 3 - Alirocumab 75 mg Q4W: <50 kg | Cohort 3 - Alirocumab 150 mg Q4W: >=50 kg | Cohort 4 - Alirocumab 150 mg Q4W: <50 kg | Cohort 4 - Alirocumab 300 mg Q4W: >=50 kg
Number analyzed (Participants) | 4 | 6 | 4 | 6 | 6 | 5 | 6 | 5
percent change | -0.4 (19.6) | -4.0 (16.0) | -7.4 (28.4) | 14.5 (19.0) | 19.3 (16.0) | -3.1 (17.5) | -32.1 (16.0) | -7.1 (17.5)

11. Secondary Outcome: Percent Change From Baseline in High Density Lipoprotein Cholesterol (HDL-C) at Week 8
Description: as for outcome 8
Time Frame: Baseline, Week 8
Population: Analysis was performed on mITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Cohort 1 - Alirocumab 30 mg Q2W: <50 kg | Cohort 1 - Alirocumab 50 mg Q2W: >=50 kg | Cohort 2 - Alirocumab 40 mg Q2W: <50 kg | Cohort 2 - Alirocumab 75 mg Q2W: >=50 kg | Cohort 3 - Alirocumab 75 mg Q4W: <50 kg | Cohort 3 - Alirocumab 150 mg Q4W: >=50 kg | Cohort 4 - Alirocumab 150 mg Q4W: <50 kg | Cohort 4 - Alirocumab 300 mg Q4W: >=50 kg
Number analyzed (Participants) | 4 | 6 | 4 | 6 | 6 | 5 | 6 | 5
percent change | 9.7 (7.1) | 16.5 (5.8) | 14.7 (7.7) | 10.6 (6.1) | 5.2 (5.8) | 13.8 (6.4) | 4.5 (5.8) | 2.8 (6.4)

12. Secondary Outcome: Percent Change From Baseline in Apolipoprotein A-1 at Week 8
Description: as for outcome 8
Time Frame: Baseline, Week 8
Population: Analysis was performed on mITT population. Here, overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Cohort 1 - Alirocumab 30 mg Q2W: <50 kg | Cohort 1 - Alirocumab 50 mg Q2W: >=50 kg | Cohort 2 - Alirocumab 40 mg Q2W: <50 kg | Cohort 2 - Alirocumab 75 mg Q2W: >=50 kg | Cohort 3 - Alirocumab 75 mg Q4W: <50 kg | Cohort 3 - Alirocumab 150 mg Q4W: >=50 kg | Cohort 4 - Alirocumab 150 mg Q4W: <50 kg | Cohort 4 - Alirocumab 300 mg Q4W: >=50 kg
Number analyzed (Participants) | 3 | 6 | 3 | 5 | 6 | 5 | 6 | 5
percent change | 4.4 (7.2) | 14.8 (5.1) | 10.7 (7.2) | 1.8 (5.6) | 8.9 (5.1) | 7.4 (5.6) | 5.8 (5.1) | 7.2 (5.6)

13. Secondary Outcome: Absolute Change From Baseline in Apolipoprotein B at Week 8
Description: as for outcome 8
Time Frame: Baseline, Week 8
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Cohort 1 - Alirocumab 30 mg Q2W: <50 kg | Cohort 1 - Alirocumab 50 mg Q2W: >=50 kg | Cohort 2 - Alirocumab 40 mg Q2W: <50 kg | Cohort 2 - Alirocumab 75 mg Q2W: >=50 kg | Cohort 3 - Alirocumab 75 mg Q4W: <50 kg | Cohort 3 - Alirocumab 150 mg Q4W: >=50 kg | Cohort 4 - Alirocumab 150 mg Q4W: <50 kg | Cohort 4 - Alirocumab 300 mg Q4W: >=50 kg
Number analyzed (Participants) | 3 | 6 | 3 | 5 | 6 | 5 | 6 | 5
mg/dL | -51.7 (15.8) | -18.5 (11.1) | -35.3 (15.8) | -53.4 (12.2) | -15.3 (11.1) | -5.4 (12.2) | -34.2 (11.1) | -63.5 (12.2)

14. Secondary Outcome: Absolute Change From Baseline in Non-High-Density Lipoprotein (Non-HDL-C) at Week 8
Description: as for outcome 8
Time Frame: Baseline, Week 8
Population: Analysis was performed on mITT population.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Cohort 1 - Alirocumab 30 mg Q2W: <50 kg | Cohort 1 - Alirocumab 50 mg Q2W: >=50 kg | Cohort 2 - Alirocumab 40 mg Q2W: <50 kg | Cohort 2 - Alirocumab 75 mg Q2W: >=50 kg | Cohort 3 - Alirocumab 75 mg Q4W: <50 kg | Cohort 3 - Alirocumab 150 mg Q4W: >=50 kg | Cohort 4 - Alirocumab 150 mg Q4W: <50 kg | Cohort 4 - Alirocumab 300 mg Q4W: >=50 kg
Number analyzed (Participants) | 4 | 6 | 4 | 6 | 6 | 5 | 6 | 5
mg/dL | -86.1 (20.8) | -28.7 (17.0) | -62.7 (22.1) | -88.5 (17.6) | -29.5 (17.0) | -0.6 (18.6) | -63.1 (17.0) | -106.4 (18.6)

15. Secondary Outcome: Absolute Change From Baseline in Total Cholesterol (Total-C) at Week 8
Description: as for outcome 8
Time Frame: Baseline, Week 8
Population: Analysis was performed on mITT population.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Cohort 1 - Alirocumab 30 mg Q2W: <50 kg | Cohort 1 - Alirocumab 50 mg Q2W: >=50 kg | Cohort 2 - Alirocumab 40 mg Q2W: <50 kg | Cohort 2 - Alirocumab 75 mg Q2W: >=50 kg | Cohort 3 - Alirocumab 75 mg Q4W: <50 kg | Cohort 3 - Alirocumab 150 mg Q4W: >=50 kg | Cohort 4 - Alirocumab 150 mg Q4W: <50 kg | Cohort 4 - Alirocumab 300 mg Q4W: >=50 kg
Number analyzed (Participants) | 4 | 6 | 4 | 6 | 6 | 5 | 6 | 5
mg/dL | -80.1 (21.4) | -20.8 (17.5) | -57.1 (22.8) | -84.4 (18.1) | -27.2 (17.5) | 5.3 (19.1) | -60.7 (17.5) | -105.1 (19.1)

16. Secondary Outcome: Absolute Change From Baseline in Lipoprotein(a) at Week 8
Description: as for outcome 10
Time Frame: Baseline, Week 8
Population: Analysis was performed on mITT population.
Measure: Least Squares Mean (Standard Error); unit: gram/Liter (g/L)
Arm/Group | Cohort 1 - Alirocumab 30 mg Q2W: <50 kg | Cohort 1 - Alirocumab 50 mg Q2W: >=50 kg | Cohort 2 - Alirocumab 40 mg Q2W: <50 kg | Cohort 2 - Alirocumab 75 mg Q2W: >=50 kg | Cohort 3 - Alirocumab 75 mg Q4W: <50 kg | Cohort 3 - Alirocumab 150 mg Q4W: >=50 kg | Cohort 4 - Alirocumab 150 mg Q4W: <50 kg | Cohort 4 - Alirocumab 300 mg Q4W: >=50 kg
Number analyzed (Participants) | 4 | 6 | 4 | 6 | 6 | 5 | 6 | 5
gram/Liter (g/L) | 0.003 (0.022) | -0.021 (0.017) | 0.007 (0.073) | -0.025 (0.020) | 0.023 (0.018) | -0.031 (0.019) | -0.002 (0.017) | -0.120 (0.020)

17. Secondary Outcome: Absolute Change From Baseline in HDL-C at Week 8
Description: as for outcome 8
Time Frame: Baseline, Week 8
Population: Analysis was performed on mITT population.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Cohort 1 - Alirocumab 30 mg Q2W: <50 kg | Cohort 1 - Alirocumab 50 mg Q2W: >=50 kg | Cohort 2 - Alirocumab 40 mg Q2W: <50 kg | Cohort 2 - Alirocumab 75 mg Q2W: >=50 kg | Cohort 3 - Alirocumab 75 mg Q4W: <50 kg | Cohort 3 - Alirocumab 150 mg Q4W: >=50 kg | Cohort 4 - Alirocumab 150 mg Q4W: <50 kg | Cohort 4 - Alirocumab 300 mg Q4W: >=50 kg
Number analyzed (Participants) | 4 | 6 | 4 | 6 | 6 | 5 | 6 | 5
mg/dL | 5.9 (3.4) | 7.7 (2.8) | 5.5 (3.7) | 4.9 (2.9) | 2.4 (2.8) | 5.9 (3.1) | 2.2 (2.8) | 1.2 (3.1)

18. Secondary Outcome: Absolute Change From Baseline in Fasting Triglyceride at Week 8
Description: as for outcome 10
Time Frame: Baseline, Week 8
Population: Analysis was performed on mITT population.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Cohort 1 - Alirocumab 30 mg Q2W: <50 kg | Cohort 1 - Alirocumab 50 mg Q2W: >=50 kg | Cohort 2 - Alirocumab 40 mg Q2W: <50 kg | Cohort 2 - Alirocumab 75 mg Q2W: >=50 kg | Cohort 3 - Alirocumab 75 mg Q4W: <50 kg | Cohort 3 - Alirocumab 150 mg Q4W: >=50 kg | Cohort 4 - Alirocumab 150 mg Q4W: <50 kg | Cohort 4 - Alirocumab 300 mg Q4W: >=50 kg
Number analyzed (Participants) | 4 | 6 | 4 | 6 | 6 | 5 | 6 | 5
mmol/L | -0.121 (0.193) | -0.076 (0.157) | 0.168 (0.226) | 0.111 (0.188) | 0.117 (0.157) | -0.045 (0.172) | -0.402 (0.157) | -0.107 (0.172)

19. Secondary Outcome: Absolute Change From Baseline in Apolipoprotein A-1 at Week 8
Description: as for outcome 8
Time Frame: Baseline, Week 8
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Cohort 1 - Alirocumab 30 mg Q2W: <50 kg | Cohort 1 - Alirocumab 50 mg Q2W: >=50 kg | Cohort 2 - Alirocumab 40 mg Q2W: <50 kg | Cohort 2 - Alirocumab 75 mg Q2W: >=50 kg | Cohort 3 - Alirocumab 75 mg Q4W: <50 kg | Cohort 3 - Alirocumab 150 mg Q4W: >=50 kg | Cohort 4 - Alirocumab 150 mg Q4W: <50 kg | Cohort 4 - Alirocumab 300 mg Q4W: >=50 kg
Number analyzed (Participants) | 3 | 6 | 3 | 5 | 6 | 5 | 6 | 5
mg/dL | 4.0 (9.3) | 17.7 (6.5) | 11.3 (9.3) | -0.4 (7.2) | 10.5 (6.5) | 8.0 (7.2) | 7.5 (6.5) | 11.0 (7.2)

20. Secondary Outcome: Absolute Change From Baseline in Ratio Apolipoprotein B/Apolipoprotein A-1 at Week 8
Description: as for outcome 8
Time Frame: Baseline, Week 8
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: ratio (Apo B/Apo A-1)
Groups:
- Cohort 3 - Alirocumab 75 mg Q4W: <50 kg: Participants with body weight < 50 kg received SC injection of alirocumab 75 mg administered Q4W up to Week 8 added to LMT.
Arm/Group | Cohort 1 - Alirocumab 30 mg Q2W: <50 kg | Cohort 1 - Alirocumab 50 mg Q2W: >=50 kg | Cohort 2 - Alirocumab 40 mg Q2W: <50 kg | Cohort 2 - Alirocumab 75 mg Q2W: >=50 kg | Cohort 3 - Alirocumab 75 mg Q4W: <50 kg | Cohort 3 - Alirocumab 150 mg Q4W: >=50 kg | Cohort 4 - Alirocumab 150 mg Q4W: <50 kg | Cohort 4 - Alirocumab 300 mg Q4W: >=50 kg
Number analyzed (Participants) | 3 | 6 | 3 | 5 | 6 | 5 | 6 | 5
ratio (Apo B/Apo A-1) | -0.363 (0.123) | -0.262 (0.087) | -0.370 (0.123) | -0.402 (0.096) | -0.190 (0.087) | -0.086 (0.096) | -0.282 (0.087) | -0.473 (0.096)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from the time of first dose of IMP up to the end of study (Week 152) regardless of seriousness or relationship to investigational product.
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'treatment emergent period' (the time from the first dose of study drug up to the last dose of study drug +70 days). Participants from Cohorts 1, 2 and 3 had an option to switch to cohort 2 dosage according to their weight category. 7 participants from Cohort 1 and 11 participants from Cohort 2 and 3 switched the dosage. Analysis was performed on safety population.
Groups:
- Cohort 1 - Alirocumab 30 mg Q2W: <50 kg: Participants with body weight < 50 kg received SC injection of alirocumab 30 mg administered Q2W up to the switch of dosage added to LMT.
- Cohort 1 - Alirocumab 50 mg Q2W: >=50 kg: Participants with body weight >= 50 kg received SC injection of alirocumab 50 mg administered Q2W up to the switch of dosage added to LMT.
- Cohort 2 - Alirocumab 40 mg Q2W: <50 kg: Participants with body weight < 50 kg received SC injection of alirocumab 40 mg administered Q2W up to the switch of dosage added to LMT.
- Cohort 2 - Alirocumab 75 mg Q2W: >=50 kg: Participants with body weight >= 50 kg received SC injection of alirocumab 75 mg administered Q2W up to the switch of dosage added to LMT.
- Cohort 3 - Alirocumab 75 mg Q4W: <50 kg: Participants with body weight < 50 kg received SC injection of alirocumab 75 mg administered Q4W up to the switch of dosage added to LMT.
- Cohort 3 - Alirocumab 150 mg Q4W: >=50 kg: Participants with body weight >= 50 kg received SC injection of alirocumab 150 mg administered Q4W up to the switch of dosage added to LMT.
- Cohort 4 - Alirocumab 150 mg Q4W: <50 kg: Participants with body weight < 50 kg received SC injection of alirocumab 150 mg administered Q4W up to the end of the OLE period (up to 130 weeks) added to LMT.
- Cohort 4 - Alirocumab 300 mg Q4W: >=50 kg: Participants with body weight >= 50 kg received SC injection of alirocumab 300 mg administered Q4W up to the end of the OLE period (up to 130 weeks) added to LMT.
- Alirocumab 40 Q2W Post-switch: Participants with body weight < 50 kg from cohort 1, 2 and 3 switched to dosage and received SC injection of alirocumab 40 mg administered Q2W from the switch up to the end of the OLE period (up to 130 weeks) added to LMT.
- Alirocumab 75 Q2W Post-switch: Participants from Cohort 1 (7 participants), Cohort 2 and Cohort 3 (11 participants) switched to dosage and received SC injection of alirocumab 75 mg administered Q2W up to the end of the OLE period (up to 130 weeks) added to LMT.
Arm/Group | Cohort 1 - Alirocumab 30 mg Q2W: <50 kg | Cohort 1 - Alirocumab 50 mg Q2W: >=50 kg | Cohort 2 - Alirocumab 40 mg Q2W: <50 kg | Cohort 2 - Alirocumab 75 mg Q2W: >=50 kg | Cohort 3 - Alirocumab 75 mg Q4W: <50 kg | Cohort 3 - Alirocumab 150 mg Q4W: >=50 kg | Cohort 4 - Alirocumab 150 mg Q4W: <50 kg | Cohort 4 - Alirocumab 300 mg Q4W: >=50 kg | Alirocumab 40 Q2W Post-switch | Alirocumab 75 Q2W Post-switch
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/6 | 0/4 | 0/6 | 0/6 | 0/5 | 0/6 | 0/5 | 0/10 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/6 | 0/4 | 0/6 | 0/6 | 0/5 | 0/6 | 0/5 | 0/10 | 0/18
Other Adverse Events (participants affected / at risk) | 4/4 | 5/6 | 1/4 | 4/6 | 5/6 | 3/5 | 3/6 | 4/5 | 7/10 | 9/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - Alirocumab 30 mg Q2W: <50 kg (N=4) | Cohort 1 - Alirocumab 50 mg Q2W: >=50 kg (N=6) | Cohort 2 - Alirocumab 40 mg Q2W: <50 kg (N=4) | Cohort 2 - Alirocumab 75 mg Q2W: >=50 kg (N=6) | Cohort 3 - Alirocumab 75 mg Q4W: <50 kg (N=6) | Cohort 3 - Alirocumab 150 mg Q4W: >=50 kg (N=5) | Cohort 4 - Alirocumab 150 mg Q4W: <50 kg (N=6) | Cohort 4 - Alirocumab 300 mg Q4W: >=50 kg (N=5) | Alirocumab 40 Q2W Post-switch (N=10) | Alirocumab 75 Q2W Post-switch (N=18)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Excessive Eye Blinking (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza Like Illness (General disorders) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Injection Site Reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Food Allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess Limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cytomegalovirus Hepatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (2)
Infectious Mononucleosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (5) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Otitis Externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Otitis Media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis Streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post Procedural Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal Mycotic Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Animal Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod Bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament Sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Post-Traumatic Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Follicle Stimulating Hormone Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Luteinising Hormone Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Low Density Lipoprotein Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 1 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyogenic Granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thoracic Outlet Syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alcohol Abuse (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depressed Mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Premenstrual Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pallor (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2017-12-11): https://cdn.clinicaltrials.gov/large-docs/92/NCT02890992/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/92/NCT02890992/SAP_001.pdf